CLINICAL TRIAL: NCT05534984
Title: A Randomized, Placebo-Controlled, Double-Blinded Trial of the Safety and Efficacy of Tecovirimat for the Treatment of Human Mpox Virus Disease
Brief Title: Study of Tecovirimat for Human Mpox Virus
Acronym: STOMP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommendation due to statistical futility
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: SIGA Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5418; 38982 (Other: DAIDS-ES ID)
Record Dates: First submitted 2022-09-08; First posted 2022-09-10 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: MPOX
Keywords: HMPXV
MeSH Terms: conditions — Mpox, Monkeypox | interventions — tecovirimat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tecovirimat (Arm A) (Experimental): Participants randomized to tecovirimat.
  Interventions: Drug: Tecovirimat Oral Capsule
- Placebo (Arm B) (Placebo Comparator): Participants randomized to placebo.
  Interventions: Drug: Placebo for Tecovirimat
- Open-Label Tecovirimat (Arm C) (Experimental): Participants assigned to open-label tecovirimat.
  Interventions: Drug: Tecovirimat Oral Capsule (Open Label)

INTERVENTIONS:
Drug: Tecovirimat Oral Capsule — * Participants weighing 25 kg to less than 40 kg - Tecovirimat 400 mg every 12 hours for 14 days
  * Participants weighing 40 kg to less than 120 kg - Tecovirimat 600 mg every 12 hours for 14 days
  * Participants weighing 120 kg and over - Tecovirimat 600 mg every 8 hours for 14 days
  Arms: Tecovirimat (Arm A)
Drug: Placebo for Tecovirimat — * Participants weighing 25 kg to less than 40 kg - Placebo for Tecovirimat 400 mg every 12 hours for 14 days
  * Participants weighing 40 kg to less than 120 kg - Placebo for Tecovirimat 600 mg every 12 hours for 14 days
  * Participants weighing 120 kg and over - Placebo for Tecovirimat 600 mg every 8 hours for 14 days
  Arms: Placebo (Arm B)
Drug: Tecovirimat Oral Capsule (Open Label) — * Participants weighing <3 kg - Tecovirimat 33.3 mg every 12 hours for 14 days
  * Participants weighing 3 kg to less than 6 kg- Tecovirimat 50 mg every 12 hours for 14 days
  * Participants weighing 6 kg to less than 13 kg - Tecovirimat 100 mg every 12 hours for 14 days
  * Participants weighing 13 kg to less than 25 kg - Tecovirimat 200 mg every 12 hours for 14 days
  * Participants weighing 25 kg to less than 40 kg - Tecovirimat 400 mg every 12 hours for 14 days
  * Participants weighing 40 kg to less than 120 kg - Tecovirimat 600 mg every 12 hours for 14 days
  * Participants weighing 120 kg and over - Tecovirimat 600 mg every 8 hours for 14 days
  Arms: Open-Label Tecovirimat (Arm C)

SUMMARY:
The purpose of this study was to see if tecovirimat is safe and successful at treating mpox. The main questions were whether tecovirimat reduced time to lesion resolution and pain compared to placebo (no treatment).

DETAILED DESCRIPTION:
This phase 3, randomized, placebo-controlled, double-blind clinical trial evaluated the efficacy of tecovirimat for the treatment of mpox. Participants who had or were at higher risk for severe disease because of their age or medical history, were pregnant or breastfeeding, or were taking medications that could have decreased their exposure to tecovirimat were assigned to receive open-label tecovirimat for 14 days. All other participants were randomized 2:1 to receive either tecovirimat or placebo for 14 days.

Randomized participants who reported severe pain 5 days after randomization (on Day 6) or later or progressed to severe disease stopped blinded study treatment and started a 14-day course of open-label tecovirimat.

Participants self-monitored lesions daily through 28 days (Day 29) or resolution, whichever came first, and completed a daily pain scale and symptom diary. Study visits occurred weekly through 28 days (Day 29) and included safety and skin assessments and specimen collections. A final study visit occurred at 56 days (Day 57) to assess for recrudescence of infection (development of new lesions after initial resolution of disease).

Version 3 of the protocol gave participants the option to enroll and complete study visits remotely. Participants did not provide specimens at remote visits.

On November 26, 2024, the Data and Safety Monitoring Board (DSMB) recommended that the study close due to statistical futility. The study team and sponsor agreed with the DSMB's recommendation and the study closed to accrual on November 27, 2024. The primary analysis report forming the basis of the primary manuscript used data from follow-up visits occurring through October 23, 2024, the data cutoff for the November 2024 DSMB review (the primary completion date). Outcome measures submitted to clinicaltrials.gov were also based on data from follow-up visits occurring through October 23, 2024, and summaries of participant flow, baseline characteristics, and adverse events submitted to clinicaltrials.gov were based on data from follow-up visits occurring through February 22, 2025 (the study completion date).

ELIGIBILITY:
Inclusion Criteria (All participants; Arms A, B, and C):

1. Laboratory-confirmed or presumptive human mpox virus (HMPXV) infection.
2. HMPXV illness of <14 days duration immediately prior to study entry.
3. At least one active (not yet scabbed) skin lesion, mouth lesion, or proctitis with or without visible ulcers.
4. Non-pregnant people of reproductive potential must agree to use at least one effective means of contraception when engaging in sexual activities that can result in pregnancy, from the time of enrollment through the end of study participation.
5. Ability to provide informed consent (for those above the legal age of consent and those providing consent for minors) and assent (for those who have reached the age of assent, but not the legal age of consent), as allowed by local ethics committees.
6. For participants to be enrolled/followed remotely, ability and willingness to participate in remote telehealth assessments (i.e., video visits).

Additional Inclusion Criteria for Arms A and B:

1. Age ≥18 years at the time of study entry.

Additional Inclusion Criteria for Arm C:

Participants who meet the above entry criteria who also meet any of the following criteria will be registered to Arm C.

1. Age <18 years at the time of study entry.
2. Those with severe HMPXV disease defined as having one or more of the following conditions:

   * Suspected or confirmed ocular involvement
   * Facial lesions on the malar, nose, or eyelid region
   * Confluent facial lesions
   * Hospitalization due to HMPXV infection or its complications
   * Lesions that require surgical intervention including debridement, urinary catheterization or sigmoidoscopy, or lesions extending below the dermis.

Those with or without severe disease and with one or more of the following:

* Severe immunosuppression
* Active skin conditions placing the person at higher risk for disseminated infection
* Breastfeeding
* Pregnancy
* Receipt of potent inducers
* Current or planned use of another investigational drug at any point during tecovirimat/placebo dosing that would be predicted to have a significant drug-drug interaction with tecovirimat therapeutics.

Exclusion Criteria (All participants; Arms A, B, and C):

1. Prior or concomitant receipt of tecovirimat (e.g., under an alternative access mechanism.
2. Planned initiation of intramuscular cabotegravir/rilpivirine during study drug administration or for two weeks following completion of study drug administration. Participants who were stable on long-acting intramuscular cabotegravir/rilpivirine were allowed to enroll.
3. Participants who, in the judgement of the investigator, will be at significantly increased risk as a result of participation in the study.
4. Participants who require intravenous dosing of tecovirimat.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilkin, MD, MPH, Study Chair — Cornell
Locations (54):
- United States (44):
  - Alabama CRS, Birmingham, Alabama
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles LGBT Center CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - University of California, Davis CRS, Sacramento, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - Harbor University of California Los Angeles Center, Torrance, California
  - University of Colorado Denver NICHD CRS, Aurora, Colorado
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - University of Miami / Jackson Memorial Hospital, Miami, Florida
  - Univ. of South Florida (USF) College of Medicine A, Tampa, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Rush University Cook County Hospital Chicago NICHD CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics, Boston, Massachusetts
  - Henry Ford Hospital CRS, Detroit, Michigan
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Mount Sinai West Samuels CRS, New York, New York
  - Harlem Prevention Center, New York, New York
  - Columbia Physicians & Surgeons (P&S) CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - Bronx-Lebanon Hospital Center NICHD CRS, New York, New York
  - Infectious Disease Clinical and Translational Research, New York, New York
  - University of Rochester Adult HIV Therapeutic, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Duke University Medical Center CRS, Durham, North Carolina
  - Wake Forest Baptist Medical Center CRS, Winston-Salem, North Carolina
  - Cincinnati CRS, Cincinnati, Ohio
  - Case Western Reserve University CTU, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital ATN CRS, Memphis, Tennessee
  - North Texas Infectious Disease Consultants, Dallas, Texas
  - UT Southwestern Infectious Disease Research Unit, Dallas, Texas
  - Houston AIDS Research Team (HART) CRS, Houston, Texas
  - University of Washington Positive Research, Seattle, Washington
- Fundacion Huesped CRS, Buenos Aires, Argentina
- Centro de Pesquisas Clínicas IC-HCFMUSP CRS, São Paulo, Brazil
- Nutricion Mexico CRS, Mexico City, Mexico
- Peru (5):
  - Centro de Investigaciones Tecnológicas, Biomédicas y Medioambientales CRS (CITBM) - Unidad de Ensayos Clínicos (UNIDEC) CRS, Callao
  - Barranco CRS, Lima
  - San Miguel CRS, Lima
  - Socios En Salud Sucursal Peru, Lima
  - Via Libre CRS, Lima
- Thailand (2):
  - Thai Red Cross AIDS Research Centre, Bangkok
  - Vaccine Trial Centre, Mahidol University CRS, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the Advancing Clinical Therapeutics Globally (ACTG) by NIH
Access Criteria: With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG.
  For what types of analyses? To achieve aims in the proposal approved by the ACTG.
  By what mechanism will data be made available? Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data

REFERENCES:
- [Derived] Chenchula S, Atal S, Ghanta MK, Uppugunduri CR, Karunakaran S, Amerneni KC, Sarma P, Prakash S, Amerneni LS, Padmavathi R, Anitha K, Sri Varshini T, Vishnu Vardhan K, Kaore S, Sadasivam B. Emerging variants of Mpox virus and tecovirimat resistance: Genomic insights and implications for treatment strategies. Virology. 2025 Jul;608:110532. doi: 10.1016/j.virol.2025.110532. Epub 2025 Apr 12. PMID 40245474
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: DAIDS EAE Manual, Version 2.0 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 58 clinical research sites in 7 countries (United States, Peru, Mexico, Thailand, Argentina, Japan, and Brazil) from September 2022 to November 2024.
Groups:
- Tecovirimat (Arm A): Participants randomized to tecovirimat.
  Tecovirimat Oral Capsule:
  * Participants weighing 25 kg to less than 40 kg - Tecovirimat 400 mg every 12 hours for 14 days
  * Participants weighing 40 kg to less than 120 kg - Tecovirimat 600 mg every 12 hours for 14 days
  * Participants weighing 120 kg and over - Tecovirimat 600 mg every 8 hours for 14 days
- Placebo (Arm B): Participants randomized to placebo.
  Placebo for Tecovirimat:
  * Participants weighing 25 kg to less than 40 kg - Placebo for Tecovirimat 400 mg every 12 hours for 14 days
  * Participants weighing 40 kg to less than 120 kg - Placebo for Tecovirimat 600 mg every 12 hours for 14 days
  * Participants weighing 120 kg and over - Placebo for Tecovirimat 600 mg every 8 hours for 14 days
- Open-Label Tecovirimat (Arm C): Participants assigned to open-label tecovirimat.
  Tecovirimat Oral Capsule (Open Label):
  * Participants weighing <3 kg - Tecovirimat 33.3 mg every 12 hours for 14 days
  * Participants weighing 3 kg to less than 6 kg- Tecovirimat 50 mg every 12 hours for 14 days
  * Participants weighing 6 kg to less than 13 kg - Tecovirimat 100 mg every 12 hours for 14 days
  * Participants weighing 13 kg to less than 25 kg - Tecovirimat 200 mg every 12 hours for 14 days
  * Participants weighing 25 kg to less than 40 kg - Tecovirimat 400 mg every 12 hours for 14 days
  * Participants weighing 40 kg to less than 120 kg - Tecovirimat 600 mg every 12 hours for 14 days
  * Participants weighing 120 kg and over - Tecovirimat 600 mg every 8 hours for 14 days
Period: Overall Study
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Started | 290 | 148 | 281
Started Treatment | 290 | 146 | 281
Started Open-Label Tecovirimat | 23 | 13 | 281
Completed | 231 | 112 | 233
Not Completed | 59 | 36 | 48
Not completed — Negative for HMPXV | 30 | 21 | 20
Not completed — Lost to Follow-up | 23 | 11 | 26
Not completed — Withdrawal by Subject | 6 | 3 | 2
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants. One participant randomized to the placebo arm was later found ineligible for study participation and excluded from all analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C) | Total
Number analyzed (Participants) | 290 | 147 | 281 | 718
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [28 to 40] | 34 [29 to 41] | 35 [30 to 41] | 34 [28 to 41]
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 214 | 103 | 194 | 511
  >=40 years | 76 | 44 | 87 | 207
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender | 284 | 141 | 269 | 694
  Transgender spectrum | 6 | 6 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 12 | 21
  Male | 286 | 142 | 269 | 697
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 137 | 60 | 133 | 330
  Not Hispanic or Latino | 150 | 82 | 143 | 375
  Unknown or Not Reported | 3 | 5 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 149 | 86 | 150 | 385
  Black or African American | 35 | 11 | 69 | 115
  Asian | 19 | 16 | 12 | 47
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 3
  American Indian or Alaska Native | 3 | 0 | 1 | 4
  Other | 28 | 11 | 15 | 54
  Multiple | 6 | 3 | 7 | 16
  Unknown | 48 | 20 | 26 | 94
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 3 | 2 | 3 | 8
  United States | 234 | 120 | 241 | 595
  Japan | 1 | 1 | 2 | 4
  Brazil | 1 | 0 | 13 | 14
  Mexico | 13 | 7 | 8 | 28
  Thailand | 10 | 4 | 7 | 21
  Peru | 28 | 13 | 7 | 48
Days from Symptom Onset, Continuous [Median (Inter-Quartile Range); unit: days] | 7 [5 to 10] | 8 [5 to 10] | 8 [6 to 10] | 8 [5 to 10]
Days from Symptom Onset, Categorical [Count of Participants; unit: Participants]
  <=5 days | 76 | 40 | 69 | 185
  >5 days | 214 | 107 | 212 | 533
Pain Level, Continuous [Median (Inter-Quartile Range); unit: score on a scale] — Pain measured on 11-point numerical rating scale where 0 = no pain and 10 = worst possible pain.
  score on a scale | 5 [2 to 7] | 5 [3 to 7] | 6 [4 to 8] | 6 [3 to 8]
Pain Level, Categorical [Count of Participants; unit: Participants]
  Mild (0-3) | 107 | 46 | 60 | 213
  Moderate (4-6) | 77 | 56 | 85 | 218
  Severe (7-10) | 106 | 45 | 136 | 287
Number of Lesions, Continuous [Median (Inter-Quartile Range); unit: lesions] | 10 [4 to 20] | 8 [3 to 17] | 30 [15 to 66] | 14 [6 to 32]
Number of Lesions, Categorical [Count of Participants; unit: Participants]
  <10 | 145 | 82 | 43 | 270
  10-100 | 139 | 64 | 197 | 400
  >100 | 6 | 1 | 41 | 48
Proctitis [Count of Participants; unit: Participants] — Population: Data missing for one participant assigned to the open-label tecovirimat arm because site did not perform the evaluation.
  Participants
    number analyzed (Participants) | 290 | 147 | 280 | 717
    Yes | 102 | 46 | 111 | 259
    No | 188 | 101 | 169 | 458
Receipt of >=1 Dose of Smallpox/Mpox Vaccine [Count of Participants; unit: Participants]
  Yes | 72 | 36 | 29 | 137
  No | 218 | 111 | 252 | 581
HIV Status [Count of Participants; unit: Participants] — Population: HIV status missing for one participant randomized to tecovirimat.
  Participants
    number analyzed (Participants) | 289 | 147 | 281 | 717
    Living with HIV | 103 | 42 | 134 | 279
    Not living with HIV | 182 | 100 | 137 | 419
    Probably living with HIV, based on best available information | 0 | 1 | 1 | 2
    Probably not living with HIV, based on best available information | 4 | 3 | 6 | 13
    No test results available | 0 | 1 | 3 | 4
Pregnant [Count of Participants; unit: Participants] — Participants who were pregnant at baseline were assigned to the open-label tecovirimat arm.
  Participants
    Yes | 0 | 0 | 1 | 1
    No | 290 | 147 | 280 | 717
Breastfeeding [Count of Participants; unit: Participants] — Participants who were breastfeeding at baseline were assigned to the open-label tecovirimat arm.
  Participants
    Yes | 0 | 0 | 0 | 0
    No | 290 | 147 | 281 | 718
Prior Receipt of Tecovirimat [Count of Participants; unit: Participants] — Participants less than 18 years of age, pregnant, or breastfeeding in the open-label arm (Arm C) were allowed up to three days of tecovirimat immediately prior to study entry.
  Participants
    Yes | 0 | 0 | 0 | 0
    No | 290 | 147 | 281 | 718

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Proportion With Clinical Resolution by Day 29
Description: Clinical resolution defined as all skin lesions scabbed, desquamated, or healed, and visible mucosal lesions healed. The cumulative incidence of clinical resolution was estimated using the Aalen-Johansen estimator. The treatment effect, i.e., the subdistribution hazard ratio of tecovirimat relative to placebo, was estimated using the Fine and Gray subdistribution proportional hazards model. All-cause death, start of open-label tecovirimat due to disease progression or severe pain, and use of other antivirals with expected activity against mpox were treated as competing events. Follow-up time was censored at last contact. Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: From study entry through 28 days of follow-up (i.e., Day 29)
Population: Eligible participants with laboratory-confirmed mpox and one or more skin or visible mucosal lesions that were able to be followed to resolution according to assigned treatment arm.
Measure: Number (95% Confidence Interval); unit: cumulative proportion of participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 225 | 111 | 227
cumulative proportion of participants | 0.83 [0.77 to 0.87] | 0.84 [0.76 to 0.90] | 0.85 [0.79 to 0.90]
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Test type: Superiority; p = 0.89, Fine and Gray — Threshold for statistical significance was 0.01907. Significance level used adjusts for interim looks according to the Lan and DeMets spending function analog of the O'Brien-Fleming boundaries; Subdistribution hazard ratio = 0.98, 98.09% CI 2-sided [0.74 to 1.31] — Subdistribution hazard ratio expressed as tecovirimat relative to placebo. Nominal 98.09% confidence interval presented adjusts for interim looks according to the Lan and DeMets spending function analog of the O'Brien-Fleming boundaries

2. Secondary Outcome: Mean Time-weighted Average of Pain Intensity Difference Over 5 Days of Treatment
Description: Pain was measured on 11-point numerical rating scale (NRS) where 0 = no pain and 10 = worst possible pain.
  Pain intensity difference at ith day of treatment (i = 2, ..., 6) calculated as NRS pain score at baseline (last available pre-treatment) minus NRS pain score on ith day of treatment
  Time-weighted average of pain intensity difference over 5 days of treatment was a weighted average of the pain intensity difference from treatment day 2 to treatment day 6, where the weights were calculated as the duration in days between the ith day of treatment and the day of the previous measurement. The lowest possible value that this could have been was -10, which would have indicated an increase in pain by 10 points on average over 5 days of treatment. The highest possible value that this could have been was +10, which would have indicated a decrease in pain by 10 points on average over 5 days of treatment.
  Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Through 5 days of treatment (i.e., Treatment Day 6)
Population: Eligible participants with laboratory-confirmed mpox and severe pain (NRS 7-10) at baseline according to assigned treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 71 | 30 | 96
score on a scale | 3.2 (2.1) | 3.1 (2.0) | 3.6 (2.1)
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Test type: Superiority; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.8 to 1.0] — Treatment group difference calculated as tecovirimat minus placebo. Confidence interval estimation assumed equal variances

3. Secondary Outcome: Mean Time-weighted Average of Pain Intensity Difference Over 14 Days of Treatment
Description: Pain was measured on 11-point numerical rating scale (NRS) where 0 = no pain and 10 = worst possible pain.
  Pain intensity difference at ith day of treatment (i = 2, ..., 15) calculated as NRS pain score at baseline (last available pre-treatment) minus NRS pain score on ith day of treatment
  Time-weighted average of pain intensity difference over 14 days of treatment was a weighted average of the pain intensity difference from treatment day 2 to treatment day 15, where the weights were calculated as the duration in days between the ith day of treatment and the day of the previous measurement. The lowest possible value that this could have been was -10, which would have indicated an increase in pain by 10 points on average over 5 days of treatment. The highest possible value that this could have been was +10, which would have indicated a decrease in pain by 10 points on average over 5 days of treatment.
  Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Through 14 days of treatment (i.e., Treatment Day 15)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 72 | 31 | 100
score on a scale | 4.8 (2.2) | 4.9 (2.1) | 5.5 (2.0)
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.1 to 0.8] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants Who Developed Severe HMPXV Disease
Description: Severe HMPXV disease was defined as one or more of the following conditions: suspected or confirmed ocular involvement, facial lesions on the malar, nose, or eyelid region, confluent facial lesions, hospitalization due to HMPXV infection or its complications, or lesions that required surgical intervention including debridement, urinary catheterization, or sigmoidoscopy, or extended below the dermis.
Time Frame: From study entry through 56 days of follow-up (i.e., Day 57)
Population: Eligible participants with laboratory-confirmed mpox who did not have severe HMPXV disease at baseline according to assigned treatment arm. Participants who had severe HMPXV disease at baseline were enrolled into Arm C.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 241 | 118 | 22
Participants | 9 | 6 | 1

5. Secondary Outcome: Number of Participants With HMPXV DNA Below Limit of Detection in Skin Lesions
Description: HMPXV DNA was measured as detected or below limit of detection. Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Baseline, Days 8, 15, 22, 29, and 57
Population: Eligible participants enrolled in-person with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 179 | 84 | 191
Participants
  Baseline: number analyzed (Participants) | 142 | 70 | 172
  Baseline | 18 | 12 | 23
  Day 8: number analyzed (Participants) | 141 | 71 | 155
  Day 8 | 68 | 26 | 66
  Day 15: number analyzed (Participants) | 130 | 66 | 151
  Day 15 | 106 | 53 | 122
  Day 22: number analyzed (Participants) | 116 | 62 | 118
  Day 22 | 110 | 59 | 105
  Day 29: number analyzed (Participants) | 118 | 65 | 112
  Day 29 | 112 | 64 | 102
  Day 57: number analyzed (Participants) | 117 | 60 | 94
  Day 57 | 115 | 60 | 92
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.10, Z-test; If there were <5 events in at least one arm, comparisons used Fisher's exact test. Otherwise, comparisons used a two-sample Z-test; Risk Difference (RD) = 11.6, 95% CI 2-sided [-2.3 to 25.5] — Treatment group difference calculated as tecovirimat minus placebo. If there were <5 events in at least one arm, melded confidence intervals are presented. Otherwise, Wald confidence intervals are presented
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.84, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 1.2, 95% CI 2-sided [-10.4 to 12.9] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Number of Participants With HMPXV DNA Below Limit of Detection in Oropharynx
Description: as for outcome 5
Time Frame: Baseline, Days 8, 15, 22, 29, and 57
Population: Eligible participants enrolled in-person with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 179 | 84 | 191
Participants
  Baseline: number analyzed (Participants) | 143 | 70 | 172
  Baseline | 85 | 45 | 48
  Day 8: number analyzed (Participants) | 147 | 73 | 157
  Day 8 | 137 | 67 | 140
  Day 15: number analyzed (Participants) | 134 | 70 | 150
  Day 15 | 132 | 68 | 142
  Day 22: number analyzed (Participants) | 122 | 65 | 122
  Day 22 | 121 | 63 | 115
  Day 29: number analyzed (Participants) | 125 | 66 | 114
  Day 29 | 123 | 64 | 107
  Day 57: number analyzed (Participants) | 120 | 62 | 98
  Day 57 | 120 | 61 | 95
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.71, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 1.4, 95% CI 2-sided [-6.1 to 8.9] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.61, Fisher Exact; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 1.4, 95% CI 2-sided [-3.5 to 8.7] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Number of Participants With HMPXV DNA Below Limit of Detection in Rectum
Description: as for outcome 5
Time Frame: Baseline, Days 8, 15, 22, 29, and 57
Population: Eligible participants enrolled in-person with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 179 | 84 | 191
Participants
  Baseline: number analyzed (Participants) | 145 | 69 | 170
  Baseline | 46 | 26 | 39
  Day 8: number analyzed (Participants) | 146 | 71 | 156
  Day 8 | 108 | 48 | 91
  Day 15: number analyzed (Participants) | 137 | 69 | 148
  Day 15 | 134 | 64 | 120
  Day 22: number analyzed (Participants) | 124 | 64 | 118
  Day 22 | 124 | 63 | 103
  Day 29: number analyzed (Participants) | 126 | 65 | 113
  Day 29 | 123 | 65 | 103
  Day 57: number analyzed (Participants) | 121 | 60 | 94
  Day 57 | 120 | 60 | 88
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.34, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 6.4, 95% CI 2-sided [-6.6 to 19.4] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.12, Fisher Exact; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 5.1, 95% CI 2-sided [-1.6 to 14.2] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Number of Participants With HMPXV DNA Below Limit of Detection in Blood
Description: HMPXV DNA measured as detected or below limit of detection. Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Baseline, Days 8, 15, 22, 29, and 57
Population: Eligible participants enrolled in-person with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 179 | 84 | 191
Participants
  Baseline: number analyzed (Participants) | 168 | 78 | 173
  Baseline | 69 | 45 | 40
  Day 8: number analyzed (Participants) | 153 | 73 | 158
  Day 8 | 139 | 65 | 127
  Day 15: number analyzed (Participants) | 139 | 70 | 153
  Day 15 | 136 | 65 | 133
  Day 22: number analyzed (Participants) | 125 | 65 | 124
  Day 22 | 122 | 62 | 106
  Day 29: number analyzed (Participants) | 127 | 67 | 116
  Day 29 | 125 | 67 | 105
  Day 57: number analyzed (Participants) | 118 | 62 | 103
  Day 57 | 118 | 62 | 99
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.68, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 1.8, 95% CI 2-sided [-6.7 to 10.3] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.12, Fisher Exact; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-1.6 to 14.0] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Number of Participants With HMPXV DNA Below Limit of Detection in Vaginal Swabs
Description: as for outcome 8
Time Frame: Baseline, Days 8, 15, 22, 29, and 57
Population: Female participants enrolled in-person with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 4 | 1 | 7
Participants
  Baseline: number analyzed (Participants) | 4 | 0 | 5
  Baseline | 0 | 0 | 1
  Day 8: number analyzed (Participants) | 4 | 1 | 4
  Day 8 | 1 | 0 | 2
  Day 15: number analyzed (Participants) | 3 | 0 | 4
  Day 15 | 1 | 0 | 2
  Day 22: number analyzed (Participants) | 4 | 1 | 3
  Day 22 | 3 | 1 | 3
  Day 29: number analyzed (Participants) | 4 | 1 | 4
  Day 29 | 4 | 1 | 3
  Day 57: number analyzed (Participants) | 3 | 1 | 2
  Day 57 | 3 | 1 | 2

10. Secondary Outcome: Cumulative Proportion With Complete Lesion Healing by Day 29
Description: Complete lesion healing was defined as all lesions re-epithelialized. The cumulative incidence of complete lesion healing was estimated using the Aalen-Johansen estimator. The treatment effect, i.e., the subdistribution hazard ratio of tecovirimat relative to placebo, was estimated using the Fine and Gray subdistribution proportional hazards model. All-cause death, start of open-label tecovirimat due to disease progression or severe pain, and use of other antivirals with expected activity against mpox were treated as competing events. Follow-up time was censored at last contact. Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: From study entry through 28 days of follow-up (i.e., Day 29)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: cumulative proportion of participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 225 | 111 | 227
cumulative proportion of participants | 0.75 [0.68 to 0.80] | 0.75 [0.66 to 0.83] | 0.69 [0.62 to 0.75]
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Test type: Superiority; p = 0.82, Fine and Gray; Subdistribution hazard ratio = 0.97, 95% CI 2-sided [0.75 to 1.26] — Subdistribution hazard ratio expressed as tecovirimat relative to placebo

11. Secondary Outcome: Number of Participants With no Missed Doses (of Last Three Prescribed Doses)
Description: Since the adherence assessment was removed from protocol version 3.0, the number of participants with adherence data was expected to be small and no formal statistical comparison between treatment arms was done. Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Days 8 and 15
Population: Eligible participants who took at least one dose of tecovirimat or placebo according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 275 | 136 | 266
Participants
  Day 8: number analyzed (Participants) | 45 | 21 | 28
  Day 8: 0 missed doses | 43 | 18 | 27
  Day 8: 1 missed doses | 0 | 0 | 1
  Day 8: 2 missed doses | 1 | 2 | 0
  Day 8: 3 missed doses | 1 | 1 | 0
  Day 15: number analyzed (Participants) | 37 | 17 | 27
  Day 15: 0 missed doses | 36 | 16 | 24
  Day 15: 1 missed doses | 1 | 1 | 2
  Day 15: 2 missed doses | 0 | 0 | 1
  Day 15: 3 missed doses | 0 | 0 | 0

12. Secondary Outcome: Median Change From Baseline in EuroQol (EQ) Visual Analogue Scale (VAS) Score
Description: Participants' self-rated health measured on a visual analogue scale (VAS) where 0 = "The worst health you can imagine" and 100 = "The best health you can imagine." Change in EQ VAS score at each timepoint calculated as absolute change from baseline (last available pre-treatment). Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Days 8, 15, and 29
Population: Eligible participants with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 241 | 118 | 239
score on a scale
  Day 8: number analyzed (Participants) | 203 | 103 | 206
  Day 8 | 10 [0 to 20] | 10 [5 to 25] | 15 [5 to 30]
  Day 15: number analyzed (Participants) | 182 | 94 | 190
  Day 15 | 20 [5 to 35] | 20 [10 to 30] | 25 [10 to 40]
  Day 29: number analyzed (Participants) | 167 | 80 | 174
  Day 29 | 20 [10 to 35] | 24.5 [10 to 30] | 25 [10 to 45]
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 29; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Number of Participants Who Reported Each Level of Response on Mobility Dimension of EuroQol EQ-5D-5L Questionnaire
Description: Participants' self-reported health state within mobility dimension of the five-dimension EuroQol EQ-5D-5L questionnaire. Participants were asked to indicate their health state by selecting the most appropriate response level for them from five ordinal response levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5).
  Results were dichotomized into no problems (level 1) and any problems (levels 2, 3, 4, and 5 combined) for reporting and analysis.
  Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Baseline, Days 8, 15, and 29
Population: Eligible participants with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 241 | 118 | 239
Participants
  Baseline: number analyzed (Participants) | 227 | 114 | 224
  Baseline: No problems | 169 | 86 | 153
  Baseline: Any problems | 58 | 28 | 71
  Day 8: number analyzed (Participants) | 218 | 106 | 219
  Day 8: No problems | 197 | 98 | 180
  Day 8: Any problems | 21 | 8 | 39
  Day 15: number analyzed (Participants) | 190 | 97 | 202
  Day 15: No problems | 184 | 96 | 188
  Day 15: Any problems | 6 | 1 | 14
  Day 29: number analyzed (Participants) | 178 | 85 | 191
  Day 29: No problems | 170 | 83 | 176
  Day 29: Any problems | 8 | 2 | 15
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.52, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.021, 95% CI 2-sided [-0.043 to 0.085] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.43, Fisher Exact; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.021, 95% CI 2-sided [-0.030 to 0.061] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 29; Test type: Superiority; p = 0.51, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.021, 95% CI 2-sided [-0.044 to 0.071] — [estimate comment as in outcome 5, analysis 1]

14. Secondary Outcome: Number of Participants Who Reported Each Level of Response on Self-Care Dimension of EuroQol EQ-5D-5L Questionnaire
Description: Participants' self-reported health state within self-care dimension of five-dimension EuroQol EQ-5D-5L questionnaire. Participants were asked to indicate their health state by selecting the most appropriate response level for them from five ordinal response levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5).
  Results were dichotomized into no problems (level 1) and any problems (levels 2, 3, 4, and 5 combined) for reporting and analysis.
  Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Baseline, Days 8, 15, and 29
Population: Eligible participants with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 241 | 118 | 239
Participants
  Baseline: number analyzed (Participants) | 226 | 114 | 224
  Baseline: No problems | 177 | 86 | 170
  Baseline: Any problems | 49 | 28 | 54
  Day 8: number analyzed (Participants) | 218 | 106 | 219
  Day 8: No problems | 203 | 99 | 195
  Day 8: Any problems | 15 | 7 | 24
  Day 15: number analyzed (Participants) | 190 | 97 | 202
  Day 15: No problems | 184 | 94 | 186
  Day 15: Any problems | 6 | 3 | 16
  Day 29: number analyzed (Participants) | 178 | 85 | 191
  Day 29: No problems | 174 | 83 | 185
  Day 29: Any problems | 4 | 2 | 6
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.93, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.003, 95% CI 2-sided [-0.055 to 0.061] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 1.00, Fisher Exact; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.001, 95% CI 2-sided [-0.061 to 0.047] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 29; Test type: Superiority; p = 1.00, Fisher Exact; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = -0.001, 95% CI 2-sided [-0.063 to 0.042] — [estimate comment as in outcome 5, analysis 1]

15. Secondary Outcome: Number of Participants Who Reported Each Level of Response on Usual Activities Dimension of EuroQol EQ-5D-5L Questionnaire
Description: Participants' self-reported health state within usual activities dimension of five-dimension EuroQol EQ-5D-5L questionnaire. Participants were asked to indicate their health state by selecting the most appropriate response level for them from five ordinal response levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5).
  Results were dichotomized into no problems (level 1) and any problems (levels 2, 3, 4, and 5 combined) for reporting and analysis.
  Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Baseline, Days 8, 15, and 29
Population: Eligible participants with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 241 | 118 | 239
Participants
  Baseline: number analyzed (Participants) | 227 | 114 | 224
  Baseline: No problems | 140 | 72 | 123
  Baseline: Any problems | 87 | 42 | 101
  Day 8: number analyzed (Participants) | 218 | 106 | 219
  Day 8: No problems | 171 | 88 | 164
  Day 8: Any problems | 47 | 18 | 55
  Day 15: number analyzed (Participants) | 190 | 97 | 202
  Day 15: No problems | 179 | 93 | 176
  Day 15: Any problems | 11 | 4 | 26
  Day 29: number analyzed (Participants) | 178 | 85 | 191
  Day 29: No problems | 172 | 82 | 171
  Day 29: Any problems | 6 | 3 | 20
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.32, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.046, 95% CI 2-sided [-0.044 to 0.136] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.78, Fisher Exact; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.017, 95% CI 2-sided [-0.052 to 0.072] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 29; Test type: Superiority; p = 1.00, Fisher Exact; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = -0.002, 95% CI 2-sided [-0.071 to 0.049] — [estimate comment as in outcome 5, analysis 1]

16. Secondary Outcome: Number of Participants Who Reported Each Level of Response on Pain/Discomfort Dimension of EuroQol EQ-5D-5L Questionnaire
Description: Participants' self-reported health state within pain/discomfort dimension of five-dimension EuroQol EQ-5D-5L questionnaire. Participants were asked to indicate their health state by selecting the most appropriate response level for them from five ordinal response levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5).
  Results were dichotomized into no problems (level 1) and any problems (levels 2, 3, 4, and 5 combined) for reporting and analysis.
  Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Baseline, Days 8, 15, and 29
Population: Eligible participants with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 241 | 118 | 239
Participants
  Baseline: number analyzed (Participants) | 227 | 114 | 224
  Baseline: No problems | 41 | 15 | 23
  Baseline: Any problems | 186 | 99 | 201
  Day 8: number analyzed (Participants) | 218 | 106 | 219
  Day 8: No problems | 119 | 59 | 98
  Day 8: Any problems | 99 | 47 | 121
  Day 15: number analyzed (Participants) | 190 | 97 | 202
  Day 15: No problems | 152 | 81 | 148
  Day 15: Any problems | 38 | 16 | 54
  Day 29: number analyzed (Participants) | 178 | 85 | 191
  Day 29: No problems | 158 | 80 | 157
  Day 29: Any problems | 20 | 5 | 34
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.86, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.011, 95% CI 2-sided [-0.105 to 0.126] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.46, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.035, 95% CI 2-sided [-0.058 to 0.128] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 29; Test type: Superiority; p = 0.12, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.054, 95% CI 2-sided [-0.015 to 0.122] — [estimate comment as in outcome 5, analysis 1]

17. Secondary Outcome: Number of Participants Who Reported Each Level of Response on Anxiety/Depression Dimension of EuroQol EQ-5D-5L Questionnaire
Description: Participants' self-reported health state within anxiety/depression dimension of five-dimension EuroQol EQ-5D-5L questionnaire. Participants were asked to indicate their health state by selecting the most appropriate response level for them from five ordinal response levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5).
  Results were dichotomized into no problems (level 1) and any problems (levels 2, 3, 4, and 5 combined) for reporting and analysis.
  Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Baseline, Days 8, 15, and 29
Population: Eligible participants with laboratory-confirmed mpox according to assigned treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 241 | 118 | 239
Participants
  Baseline: number analyzed (Participants) | 227 | 114 | 224
  Baseline: No problems | 78 | 50 | 63
  Baseline: Any problems | 149 | 64 | 161
  Day 8: number analyzed (Participants) | 218 | 106 | 219
  Day 8: No problems | 121 | 59 | 114
  Day 8: Any problems | 97 | 47 | 105
  Day 15: number analyzed (Participants) | 190 | 97 | 202
  Day 15: No problems | 123 | 70 | 119
  Day 15: Any problems | 67 | 27 | 83
  Day 29: number analyzed (Participants) | 178 | 85 | 191
  Day 29: No problems | 138 | 65 | 127
  Day 29: Any problems | 40 | 20 | 64
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 8; Test type: Superiority; p = 0.98, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.002, 95% CI 2-sided [-0.114 to 0.117] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 15; Test type: Superiority; p = 0.19, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 0.074, 95% CI 2-sided [-0.038 to 0.186] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Treatment group difference at Day 29; Test type: Superiority; p = 0.85, Z-test; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = -0.011, 95% CI 2-sided [-0.120 to 0.098] — [estimate comment as in outcome 5, analysis 1]

18. Secondary Outcome: Proportion of Participants With Grade 3 or Greater Treatment-emergent Adverse Event
Description: Study protocol required reporting of all adverse events (AEs) that (1) led to a change in study treatment regardless of grade, (2) met the serious AE (SAE) or Expedited AE (EAE) reporting requirement, and (3) were Grade 3 or greater. AEs were graded using the DAIDS AE Grading Table (Version 2.1).
  Severity Grade: 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Life-Threatening, 5 = Death
  Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Through 56 days of follow-up (i.e., Day 57)
Population: Eligible participants who took at least one dose of tecovirimat or placebo according to initial treatment received. Participants enrolled after October 23, 2024 were excluded.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 275 | 136 | 266
proportion of participants | 0.044 [0.019 to 0.068] | 0.044 [0.010 to 0.079] | 0.071 [0.040 to 0.102]
Statistical Analysis 1: Comparison: Tecovirimat (Arm A) vs Placebo (Arm B); Test type: Superiority; p = 0.98, Z-test; Risk Difference (RD) = -0.000, 95% CI 2-sided [-0.043 to 0.042] — Treatment group difference calculated as tecovirimat minus placebo. Wald confidence intervals are presented

19. Secondary Outcome: Number of Participants Who Died From Any Cause
Description: Includes data from follow-up visits occurring through October 23, 2024.
Time Frame: Through 56 days of follow-up (i.e., Day 57)
Population: Eligible participants according to assigned treatment arm. Participants enrolled after October 23, 2024 were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 275 | 137 | 266
Participants | 0 | 0 | 0

20. Secondary Outcome: Tecovirimat Concentrations in Children Less Than 18 Years of Age
Description: Plasma tecovirimat concentrations were quantified using validated liquid chromatography tandem mass spectrometry (LC-MS/MS) methods. The lower limit of quantification was 5.0 ng/mL.
Time Frame: On Day 8, blood samples were collected pre-dose and at 1, 2, 3, 4, 6, 8, and 10 hours post-dose. On Day 15, a single blood sample was collected within 4 hours of study product administration.
Population: Measure was not analyzed since only one participant aged <18 years was enrolled and no aggregate results were available for posting.
Arm/Group | Tecovirimat (Arm A) | Placebo (Arm B) | Open-Label Tecovirimat (Arm C)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From study entry to study completion at Day 57 or premature study discontinuation.
Description: AEs that led to change in study treatment regardless of grade, met serious AE definition or expedited AE reporting requirement, or were Grade 3 or higher were reported and graded using DAIDS AE Grading Table (v2.1). Participants who started open-label tecovirimat were reported separately from their initial treatment arm, thus:
  at Risk (Arm A) = Started Treatment (Arm A) - Started Open-Label (Arm A)
  at Risk (Arm B) = Started Treatment (Arm B) - Started Open-Label (Arm B) - 1 ineligible
Groups:
- Tecovirimat (Arm A) to Open-Label Tecovirimat (Arm C): Participants randomized to tecovirimat who started open-label tecovirimat.
- Placebo (Arm B) to Open-Label Tecovirimat (Arm C): Participants randomized to placebo who started open-label tecovirimat.
Arm/Group | Tecovirimat (Arm A) | Tecovirimat (Arm A) to Open-Label Tecovirimat (Arm C) | Placebo (Arm B) | Placebo (Arm B) to Open-Label Tecovirimat (Arm C) | Open-Label Tecovirimat (Arm C)
All-Cause Mortality (participants affected / at risk) | 0/267 | 0/23 | 0/132 | 0/13 | 0/281
Serious Adverse Events (participants affected / at risk) | 4/267 | 2/23 | 0/132 | 2/13 | 14/281
Other Adverse Events (participants affected / at risk) | 7/267 | 12/23 | 4/132 | 9/13 | 14/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecovirimat (Arm A) (N=267) | Tecovirimat (Arm A) to Open-Label Tecovirimat (Arm C) (N=23) | Placebo (Arm B) (N=132) | Placebo (Arm B) to Open-Label Tecovirimat (Arm C) (N=13) | Open-Label Tecovirimat (Arm C) (N=281)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Monkeypox (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Proctitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecovirimat (Arm A) (N=267) | Tecovirimat (Arm A) to Open-Label Tecovirimat (Arm C) (N=23) | Placebo (Arm B) (N=132) | Placebo (Arm B) to Open-Label Tecovirimat (Arm C) (N=13) | Open-Label Tecovirimat (Arm C) (N=281)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 4 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Acute HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes simplex anorectal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Monkeypox (Infections and infestations) | 0 | 4 | 0 | 5 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Paraphimosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Penile swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Enrollment to the trial was stopped early due to statistical futility based on a recommendation from an independent DSMB at the second interim efficacy review.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (3):
  • Study Protocol and Informed Consent Form: V 3.0 (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT05534984/Prot_ICF_000.pdf
  • Study Protocol: Clarification Memo #3 07SEP2023 (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT05534984/Prot_001.pdf
  • Statistical Analysis Plan (2025-08-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT05534984/SAP_002.pdf